CLINICAL TRIAL: NCT00060931
Title: A Randomized, Double-Blind, Multicenter Study Comparing the Effects of Carvedilol and Metoprolol on Glycemic Control in Hypertensive Patients With Type II Diabetes Mellitus.
Brief Title: Effect Of Carvedilol Versus Metoprolol On Glycemic Control In Patients With Type II Diabetes And Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105517/347
Record Dates: First submitted 2003-05-15; First posted 2003-05-16 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension
Keywords: hypertension; beta-blockers; Type 2 diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carvedilol
Drug: metoprolol
  Other Names: carvedilol

SUMMARY:
Evaluation of the effect of two different antihypertensive treatments on control of glucose in Type II diabetic patients with high blood pressure

ELIGIBILITY:
Inclusion criteria:

* Patients at screening must be insulin producing Type II diabetics (C peptide positive).
* Patients must have a history of mild to moderate hypertension (140-179 systolic blood pressure; 90-1-9 diastolic blood pressure)
* Patients must be on a stable regimen of ACE (angiotensin converting enzyme) / ARB (angiotensin receptor blocker) treatment alone or in combination with other treatments.
* Patients must be on stable antidiabetic regimen (drug treated or diet alone).
* Patient''s laboratory result for HbA1c must be 6.5 - 8.5 (drug treated) or 6.5 - 7.5 (diet alone).

Exclusion criteria:

* Patients using beta-blocker therapy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2001-06; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 5 months | 5 months

SECONDARY OUTCOMES:
Blood pressure at 3 and 5 months Body weight at 3 and 5 months Lab levels (glucose, insulin, triglycerides, cholesterol, and albumin:creatinine ratio) at 3 and 5 months. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (100):
- United States (100):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Columbia, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Derby, Connecticut
  - GSK Investigational Site, Farmington, Connecticut
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Meyers, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Saint Petersberg, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, West Evanston, Illinois
  - GSK Investigational Site, Newburgh, Indiana
  - GSK Investigational Site, Wabash, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Auburn, Maine
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Ayer, Massachusetts
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Waltham, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Waterford, Michigan
  - GSK Investigational Site, Gulfport, Mississippi
  - GSK Investigational Site, Camden, New Jersey
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Linwood, New Jersey
  - GSK Investigational Site, Margate City, New Jersey
  - GSK Investigational Site, Sea Girt, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Flushing, New York
  - GSK Investigational Site, Fulton, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, Lancaster, New York
  - GSK Investigational Site, Liverpool, New York
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Scarsdale, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Tonawanda, New York
  - GSK Investigational Site, Williamsville, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Connellsville, Pennsylvania
  - GSK Investigational Site, Downington, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Fleetwood, Pennsylvania
  - GSK Investigational Site, Morrisville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Philipsburg, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, West Grove, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, White River Junction, Utah
  - GSK Investigational Site, Christiansburg, Virginia
  - GSK Investigational Site, Falls Church, Virginia
  - GSK Investigational Site, Fredericksburg, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Springfield, Virginia